CLINICAL TRIAL: NCT03389230
Title: Phase I Study of Cellular Immunotherapy Using Memory-Enriched T Cells Lentivirally Transduced to Express a HER2-Specific, Hinge-Optimized, 41BB-Costimulatory Chimeric Receptor and a Truncated CD19 for Patients With Recurrent/Refractory Malignant Glioma
Brief Title: Memory-Enriched T Cells in Treating Patients With Recurrent or Refractory Grade III-IV Glioma
Status: Active, not recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: City of Hope Medical Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 16064; NCI-2017-01755 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 16064 (Other: City of Hope Medical Center); P30CA033572 (NIH)
Record Dates: First submitted 2017-12-27; First posted 2018-01-03 (Actual); Last update posted 2026-02-04 (Actual); Status verified 2026-02

CONDITIONS: Glioblastoma; Malignant Glioma; Recurrent Glioma; Refractory Glioma; WHO Grade III Glioma
MeSH Terms: conditions — Glioblastoma; Glioma | interventions — Leukapheresis

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (3):
- Arm I (intratumoral/intracavitary delivery) (Experimental): Patients receive autologous HER2(EQ)BBzeta/CD19t+ Tcm cells via intratumoral/intracavitary catheter over 5 minutes weekly for 3 weeks. Beginning as early as 1 week later, patients may receive additional T cell infusions as long as patients remain eligible and there is product available. Patients who progress on intracavitary or intratumoral administration may move to alternative delivery routes for the optional infusions.
  Interventions: Biological: HER2(EQ)BBζ/CD19t+ T cells; Other: Laboratory Biomarker Analysis; Procedure: Leukapheresis
- Arm II (dual delivery Tcm enriched) (Experimental): Patients receive autologous HER2(EQ)BBzeta/CD19t+ Tcm cells via intratumoral/intracavitary catheter and intraventricular catheter over 5 minutes weekly for 3 weeks. Beginning as early as 1 week later, patients may receive additional T cell infusions as long as patients continue to remain eligible and there is product available. Based on clinical response after the first 3 infusions, the study principal investigator may decide to continue with the optional infusions at either one or both sites (instead of requiring injections at both sites).
  Interventions: Biological: HER2(EQ)BBζ/CD19t+ T cells; Other: Laboratory Biomarker Analysis; Procedure: Leukapheresis
- ARM III (dual delivery Tn/mem enriched) (Experimental): Patients receive autologous HER2(EQ)BBzeta/CD19t+ Tn/mem cells via intratumoral/intracavitary catheter and intraventricular catheter over 5 minutes weekly for 3 weeks. Beginning as early as 1 week later, patients may receive additional T cell infusions as long as patients continue to remain eligible and there is product available. Based on clinical response after the first 3 infusions, the study principal investigator may decide to continue with the optional infusions at either one or both sites (instead of requiring injections at both sites).
  Interventions: Biological: HER2(EQ)BBζ/CD19t+ T cells; Other: Laboratory Biomarker Analysis; Procedure: Leukapheresis

INTERVENTIONS:
Biological: HER2(EQ)BBζ/CD19t+ T cells — Given via catheter
Other: Laboratory Biomarker Analysis — Correlative studies
Procedure: Leukapheresis — Undergo leukapheresis
  Other Names: Leukocytopheresis; Therapeutic Leukopheresis

SUMMARY:
This phase I trial studies the side effects and best dose of memory-enriched T cells in treating patients with grade II-IV glioma that has come back (recurrent) or does not respond to treatment (refractory). Memory enriched T cells such as HER2(EQ)BBζ/CD19t+ T cells may enter and express its genes in immune cells. Immune cells can be engineered to kill glioma cells in the laboratory by inserting a piece of deoxyribonucleic acid (DNA) into the immune cells that allows them to recognize glioma cells. A vector called lentivirus is used to carry the piece of DNA into the immune cell. It is not known whether these immune cells will kill glioma tumor cells when given to patients.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To assess the feasibility and safety of cellular immunotherapy utilizing ex vivo expanded autologous memory-enriched T cells that are genetically modified using a self-inactivating (SIN) lentiviral vector to express a HER2-specific, hinge-optimized, 41BB-costimulatory chimeric antigen receptor (CAR), as well as a truncated human CD19 (HER2[EQ]BBzeta/CD19t+) for participants with recurrent/refractory malignant glioma in one of the following ways: Arm 1 (intracavitary/intratumoral HER2(EQ)BBzeta/CD19+ T CM), Arm 2 (dual delivery [both intracavitary/intratumoral and intraventricular] of HER2(EQ)BBzeta/CD19+ T CM), or Arm 3 (dual delivery [both intracavitary/intratumoral and intraventricular] of HER2(EQ)BBzeta/CD19+ T N/MEM).

II. To determine maximum tolerated dose schedule (MTD) and a recommended Phase II dosing plan (RP2D) for arm 3 (dual delivery).

SECONDARY OBJECTIVES:

I. To describe persistence and expansion of CAR T cells in tumor cyst fluid, peripheral blood and cerebral spinal fluid (CSF).

II. To describe cytokine levels (tumor cyst fluid, peripheral blood, and CSF) over the study period.

III. In research participants who receive the full schedule of 3 CAR T cell doses:

IIIa. To estimate median progression free survival (PFS) rate. IIIb. To estimate disease response rates. IIIc. To estimate median overall survival (OS).

IV. In research participants who continue to receive infusions after progressing:

IVa. Estimate disease response. IVb. Describe CAR T cell and endogenous immune populations, as well as cytokine and microenvironment profiles (cerebral spinal fluid [CSF], cyst fluid, peripheral blood) considering post progression therapy(ies), if applicable.

V. For study participants who undergo an additional biopsy/resection or autopsy:

Va. Evaluate CAR T cell persistence in the tumor micro-environment and the location of the CAR T cells with respect to the injection.

Vb. Evaluate HER2 antigen expression levels pre and post CAR T cell therapy.

OUTLINE: This is a dose-escalation study of autologous HER2(EQ)BBζ/CD19t+ T cells. Participants are assigned to 1 of 3 arms.

ARM I: Patients receive autologous HER2(EQ)BBzeta/CD19t+ Tcm cells via intratumoral/intracavitary catheter over 5 minutes weekly for 3 weeks. Beginning as early as 1 week later, patients may receive additional T cell infusions as long as patients remain eligible and there is product available. Patients who progress on intracavitary or intratumoral administration may move to alternative delivery routes for the optional infusions.

ARM II: Patients receive autologous HER2(EQ)BBzeta/CD19t+ Tcm cells via intratumoral/intracavitary catheter and intraventricular catheter over 5 minutes weekly for 3 weeks. Beginning as early as 1 week later, patients may receive additional T cell infusions as long as patients continue to remain eligible and there is product available. Based on clinical response after the first 3 infusions, the study principal investigator may decide to continue with the optional infusions at either one or both sites (instead of requiring injections at both sites).

ARM III: Patients receive autologous HER2(EQ)BBzeta/CD19t+ Tn/mem cells via intratumoral/intracavitary catheter and intraventricular catheter over 5 minutes weekly for 3 weeks. Beginning as early as 1 week later, patients may receive additional T cell infusions as long as patients continue to remain eligible and there is product available. Based on clinical response after the first 3 infusions, the study principal investigator may decide to continue with the optional infusions at either one or both sites (instead of requiring injections at both sites).

After completion of study treatment, patients are followed up at 4 weeks, 3, 6, 8, 10, and 12 months, then annually for at least 15 years.

ELIGIBILITY:
Inclusion Criteria:

* Participant has a prior histologically-confirmed diagnosis of a grade III or IV glioma, or has a prior histologically-confirmed diagnosis of a grade II glioma and now has radiographic progression consistent with a grade III or IV malignant glioma (MG)
* Karnofsky performance status (KPS) >= 60%
* Life expectancy > 4 weeks
* The effects of HER2(EQBBzeta/CD19t+ T cells on the developing fetus are unknown. For this reason, women of child-bearing potential and men must agree to use adequate contraception (hormonal or barrier method of birth control or abstinence) prior to study entry and for six months following duration of study participation; should a woman become pregnant or suspect that she is pregnant while participating on the trial, she should inform her treating physician immediately
* City of Hope (COH) Clinical Pathology confirms HER2+ tumor expression by immunohistochemistry (>= 20%, 1+)
* All research participants must have the ability to understand and the willingness to sign a written informed consent

  * Note: For research participants who do not speak English, a short form consent may be used with a COH certified interpreter/translator to proceed with screening and leukapheresis, while the request for a translated full consent is processed; however, the research participant is allowed to proceed with rickham placement and CAR T cell infusion only after the translated full consent form is signed
* ELIGIBILITY TO PROCEED WITH PERIPHERAL BLOOD MONONUCLEAR CELL (PBMC) COLLECTION
* Research participant must not require more than 2 mg three times daily (TID) of dexamethasone on the day of PBMC collection.
* Research participant must have appropriate venous access
* At least 2 weeks must have elapsed since the research participant received his/her last dose of prior targeted agents, chemotherapy or radiation; at the principal investigator's discretion, exception can be made for investigational agents that are delivered locally into the CSF
* ELIGIBILITY TO PROCEED WITH RICKHAM PLACEMENT

  * Once research participants meet eligibility to proceed with Rickham placement, they will be deemed accrued on to the study

    * Note: if the participant had received prior targeted radiation and new lesions have appeared outside of that targeted area, then that may be deemed radiographic evidence of measurable disease even if 12 weeks have not elapsed
* Creatinine < 1.6 mg/dL
* White blood cell (WBC) > 2,000/dl (or absolute neutrophil count [ANC] > 1,000)
* Platelets >= 100,000/dl
* International normalized ratio (INR) < 1.3
* Bilirubin < 1.5 mg/dL
* Alanine aminotransferase (ALT) and aspartate aminotransferase (AST) < 2.5 x upper limits of normal
* ELIGIBILITY TO PROCEED WITH CAR T CELL INFUSION
* Research participant has a released cryopreserved CAR T cell product
* Research participant does not require supplemental oxygen to keep saturation greater than 95% and/or does not have presence of any radiographic abnormalities on chest x-ray that are progressive
* Research participants does NOT have any known history of congestive heart failure (CHF) or cardiac symptoms consistent with NYHA classification III-IV within 6 months prior to Day 1 of protocol treatment, cardiomyopathy, myocarditis, myocardial infarction (MI), exposure to cardiotoxic medications or with clinical history suggestive of the above must have an EKG and echocardiogram (ECHO) performed within 42 days prior to registration and as clinical indicated while on treatment
* If the research participant has new symptoms of CHF, cardiomyopathy, myocarditis, MI, or exposure to cardiotoxic medications they already had a cardiac consultation, creatinine phosphokinase (CPK), and troponin testing at pre study deeming them fit for study participation
* Research participant does not have a fever exceeding 38.5 degrees Celsius (C); there is an absence of positive blood cultures for bacteria, fungus, or virus within 48-hours prior to T cell infusion and/or there aren't any indications of meningitis
* Research participant serum total bilirubin or transaminases does not exceed 2 x normal limit
* Research participant serum creatinine < 1.8 mg/dL
* Research participant does not have uncontrolled seizure activity following surgery prior to starting the first T cell dose
* Research participant platelet count must be > 100,000; however, if platelet level is between 75,000-99,000, then CAR T-cell infusion may proceed after platelet transfusion is given and the post transfusion platelet count is >= 100,000
* Research participants must not require more than 2 mg TID of dexamethasone during CAR T cell therapy
* Wash-out requirements (standard or investigational):

  * At least 6 weeks since the completion of a nitrosourea-containing chemotherapy regimen; and
  * At least 23 days must have passed since the completion of Temodar and/or 4 weeks for any other non-nitrosourea-containing cytotoxic chemotherapy regimen; if a participant's most recent treatment was with a targeted agent only, and s/he has recovered from any toxicity of this targeted agent, then a waiting period of only 2 weeks is needed from the last dose and the start of CAR T cell infusion with the exception of bevacizumab where a wash out period of at least 4 weeks is required before starting CAR T cell therapy

Exclusion Criteria:

* Research participant requires supplemental oxygen to keep saturation greater than 95% and the situation is not expected to resolve within 2 weeks
* Research participants with a known history of congestive heart failure (CHF) or cardiac symptoms consistent with New York Heart Association (NYHA) classification III-IV within 6 months prior to Day 1 of protocol treatment, cardiomyopathy, myocarditis, myocardial infarction (MI), exposure to cardiotoxic medications or with clinical history suggestive of the above must have an electrocardiogram (EKG) and echocardiogram (ECHO) performed within 42 days prior to registration and as clinically indicated while on treatment
* Research participants with new symptoms of CHF, cardiomyopathy, myocarditis, MI, or exposure to cardiotoxic medications must have a cardiac consultation, creatinine phosphokinase (CPK), and troponin testing at pre -study and as clinically indicated
* Research participant requires dialysis
* Research participant has uncontrolled seizure activity and/or clinically evident progressive encephalopathy
* Failure of research participant to understand the basic elements of the protocol and/or the risks/benefits of participating in this phase I study; a legal guardian may substitute for the research participant
* Research participants with any non-malignant intercurrent illness which is either poorly controlled with currently available treatment, or which is of such severity that the investigators deem it unwise to enter the research participant on protocol shall be ineligible
* Research participants with any other active malignancies
* Research participants being treated for severe infection or who are recovering from major surgery are ineligible until recovery is deemed complete by the investigator
* Research participants with any uncontrolled illness including ongoing or active infection; research participants with known active hepatitis B or C infection; research participants with any signs or symptoms of active infection, positive blood cultures or radiological evidence of infections
* Research participants who have confirmed human immunodeficiency virus (HIV) positivity within 4 weeks of enrollment

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 29 (Actual)
Dates: Start 2018-08-14 (Actual); Primary Completion 2026-12-29 (Estimated); Study Completion 2026-12-29 (Estimated)

PRIMARY OUTCOMES:
Incidence of grade 3 adverse events | Up to 3 years
  Tables will be created to summarize all toxicities and side effects by dose, time post treatment, organ, severity and arm.
Dose limiting toxicities (DLT) | Up to 3 years
  Rate and associated 90% Clopper and Pearson binomial confidence limits (90% confidence interval [CI]) will be estimated for participants' experiencing DLTs at the recommended phase 2 dose (RP2D) schedule.
Incidence of adverse events | Up to 3 years
  Will be graded according to Common Terminology Criteria for Adverse Events (CTCAE) version 5.0. Tables will be created to summarize all toxicities and side effects by dose, time post treatment, organ, severity and arm.

SECONDARY OUTCOMES:
Chimeric antigen receptor (CAR) T cells detected in tumor cyst fluid, peripheral blood, and cerebrospinal fluid (CSF) | Up to 3 years
  Statistical and graphical methods will be used to describe persistence and expansion of the CAR T cells (tumor cyst fluid, peripheral blood and CSF) over the study period. In study participants that undergo a second biopsy resection or following autopsy, T cells numbers, location, and antigen levels will be described.
Tumor cyst fluid, peripheral blood, and cerebrospinal fluid (CSF) cytokine levels | Up to 3 years
  Statistical and graphical methods will be used to describe persistence and expansion of cytokine levels (tumor cyst fluid, peripheral blood, and CSF) over the study period.
Progression free survival | At 6 months
  Kaplan Meier methods will be used
Overall Survival (OS) | At 6 months
  Kaplan Meier methods will be used to estimate median OS and graph the results.
Disease response | Up to 3 years
  Will be measured by Response Assessment in Neuro-Oncology Criteria (RANO) criteria. Will estimate the rate (90% CI) progression free at 6 months and rate (90% CI) with disease response.
Chimeric antigen receptor (CAR) T cells detected in tumor tissue | Up to 3 years
  T cells numbers, location, and antigen levels will be described.
HER2 antigen expression levels in tumor tissue | Up to 3 years

CONTACTS AND LOCATIONS:
Overall Officials: Behnam Badie, Principal Investigator — City of Hope Medical Center
Locations (1):
- City of Hope Medical Center, Duarte, California, United States